CLINICAL TRIAL: NCT05719766
Title: Perspective Study on How Can the Incentive Integrated E-IBD Chronic Disease Management Model Improve the Quality of Life in IBD Patients
Brief Title: Effect of Incentive Integrated E-IBD Chronic Disease Management Model on the Quality of Life in IBD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20230049
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine follow-up group (No Intervention)
- IBD Disease Management Research Group (Experimental)
  Interventions: Other: education ,psycological support and social support

INTERVENTIONS:
Other: education ,psycological support and social support — we would give targeted-education according to our patients' need(reflected via questionnaire; we would provide psycological and social support to patients based on their need reflected by questionnaire
  Arms: IBD Disease Management Research Group

SUMMARY:
This study aims to prospectively explore the effect of incentive-integrated E-IBD (electronic inflammatory bowel disease) chronic disease management model on the improvement of IBD quality of life, and provide a more effective chronic disease management model for improving the quality of life and social participation of IBD patients.The investigators firstly identify the IBD patients in need of empowerment disease activities through the questionnaire .Then, the investigators feedback the patients' education content according to their needs found.Based on the social support network of patient organization and the medical support network of tertiary medical institutions, the investigators complete the empowerment process of IBD patients' self-management initiative and self-management ability, through the internet. Finally ,the investigators evaluate the quality of life(QoL), social participation,disease self-management level via questionnaire . The primary outcome is the improvement of QoL score after three months' intervention.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinically diagnosed IBD patients,according to the criteria of the Inflammatory Bowel Group of the Gastroenterology Branch of the Chinese Medical Association in 2018;
* 2.Aged 18 to 75 years old;
* 3.Understand and comply with the requirements of the program and sign informed consent.
* 4.Identified as need intervention according to the patient identification questionnaire screening;
* 5.Patients with the ability to complete all course training and/or follow-up work;
* 6.Enrolled at least one year ahead of end of this study(for garantee of enough folllow-up time).

Exclusion Criteria:

* 1.Unable or unwilling to sign the consent form, or unable to follow the research procedure;
* 2.Patients who have had a stoma or ileorectal anastomosis (partial scales are not available);
* 3.Patients who do not complete training on time or do not complete follow-up assessments in their entirety;
* 4.Patients with other malignancies or life-threatening complications；
* 5.Pregnancy or lactation；
* 6.Patients whose remaining follow-up time less than one year before the end of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Improved score of Quality of Life after three months | three months
  Improvement score of quality of life via short inflammatory bowel disease questionnaire(SIBDQ, score scale:0~70 points) after intervention for three months,higher scores mean better quality of life.

SECONDARY OUTCOMES:
Decreased score of Socially activity limited rating | three months,one year
  Improvement score of socially activity limited rating after intervention for three months, or one year.
Decreased score of Hospital Anxiety and Depression Scale | three months,one year
  improvement score of anxiety or depression via Hospital Anxiety and Depression Scale after intervention for three months, or one year. Lower scores mean the less anxiety or depression of the patients.
Increasion of disease kownledge | three months,one year
  improvement of disease kownledge via Crohn's and Colitis Knowledge Score(CCKOWN， score scale: 0~24 points) after intervention for three months, or one year. Higher scores mean better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Yan chen, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (4):
- China (4):
  - Center of Inflammatory Bowel Disease, Department of Gastroenterology, the Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Department of Gastroenterology, Huzhou Central Hospital, Huzhou
  - Department of Gastroenterology, Ruijin Hospital, Shanghai
  - Department of Gastroenterology, Shaoxing Central Hospital, Shaoxing

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391